CLINICAL TRIAL: NCT04580810
Title: Addressing Health Disparities by Providing Evidence-Based Treatment in the Black Church
Brief Title: Black Church Treatment Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-01366; R01AA028778-01 (NIH)
Record Dates: First submitted 2020-10-07; First posted 2020-10-08 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT4CBT in the Black Church (Experimental): The 'CBT for CBT' program is modeled closely on our NIDA-published CBT manual. Seven core skill modules will cover the following topics, which correspond to the major session topics in the manual:
  Understanding and changing patterns of alcohol use, Coping with craving, Substance refusal skills, Seemingly irrelevant decisions, Planning for emergencies, and Problem-solving skills. Staying Safe
  Interventions: Behavioral: CBT4CBT in the Black Church
- Community Based Treatment as Usual (No Intervention): Treatment as usual, typically groups, offered by a specialty community based treatment center (MCCA)

INTERVENTIONS:
Behavioral: CBT4CBT in the Black Church — Use of Computer Based Treatment for Cognitive Behavioral Therapy for alcohol use disorder offered in a Black church setting
  Arms: CBT4CBT in the Black Church

SUMMARY:
This study will conduct a randomized clinical trial comparing levels of treatment initiation, engagement, and alcohol outcomes for a novel treatment strategy (CBT4CBT delivered in the Black church) compared with traditional outpatient specialty addiction treatment for a large sample of Black adults with AUD.

The purpose of this randomized clinical trial is to determine which setting (church or specialty clinic) (1) has better treatment initiation and retention rates and (2) better AUD outcomes as measured by percentage of days abstinent (PDA) (8 weeks, 3, 6 and 9 months follow up).

DETAILED DESCRIPTION:
This study is a randomized control trial focusing on rates of treatment initiation, engagement, and outcome in Black adults assigned to CBT4CBT in the Black Church relative to the standard of care for this population. This study is focusing on individuals with AUD as the needs assessment indicated that as the most common substance use problem in this setting. Moreover, our focus groups and work with Church staff has indicated that alcohol use is less stigmatized within the Black and the Church communities than other substance use. Thus, while individuals with other substance use will be included, positioning the study as focusing primarily on alcohol use will avoid potential issues of stigma and thus may facilitate recruitment.

Selecting a comparison condition for this novel intervention strategy is complex.

As the primary rationale for delivering treatment in the Black church setting is that this national network is seen as a trusted institution in the Black community, our research questions center around (1) whether delivering CBT4CBT in the Black church is a safe and effective alternative to standard care, (2) whether it engages and retains individuals better than standard specialty care, (3) the extent to which this strategy reaches individuals who would not otherwise seek treatment for AUD, (4) what kinds of individuals are particularly suited to this setting, and (5) the relative costs of this novel form of treatment delivery. Thus, a standard specialty care at Midwestern Connecticut Council on Alcohol (MCCA) as the comparison condition was selected. MCCA is a non-profit, community-based provider in the predominantly Black Dixwell neighborhood, not far from Dixwell Church and has a positive reputation in the Black community. The primary treatment modality is group therapy. In 2019, MCCA treated over 500 unique individuals (44% female, 35% African American, 20% Latino). MCCA staff are diverse and multidisciplinary. Clinic Director Steven Palma has agreed to provide a dedicated triage slot for this study so individuals can be admitted and assigned a group within one week, reducing a key barrier.

The two study settings will be balanced in several ways, with few barriers to care, both in the same neighborhood, and assignment of participants to a group within one week of randomization, thus preserving equipoise and balancing attractiveness of both sites to participants as much as possible. They will differ primarily in setting (church versus specialty care), in treatment content (CBT4CBT with spirituality elements versus group treatment with some CBT content), and group leaders (CHAs versus masters-level staff).

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* current AUD as their principal substance use disorder, confirmed via MINI100 interview, with some drinking in the past 28 days
* English-speaking

Exclusion Criteria:

* inability to provide informed consent or participate in the study procedures as proposed in the consent
* active suicidal or homicidal ideation or an unstable psychotic disorder (schizophrenia, schizoaffective disorder) or mood disorder (bipolar disorder, severe major depressive disorder),
* current engagement in substance use treatment, and
* an unwillingness to be randomized to either condition. Individuals with comorbid substance use disorders will be included, as multiple substances of use are common in this population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2025-09-05 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
Rates of treatment initiation | 8 weeks
  Rates of treatment initiation as measured by proportion of participants completing at least one session at the assigned site
Rates of engagement in treatment | 8 weeks
  Rates of engagement in treatment operationalized by proportion retained at the 4-week point at the assigned site
Percent days abstinent from alcohol | 8 weeks
  Percent days abstinent from alcohol operationalized by Timeline Follow Back

CONTACTS AND LOCATIONS:
Overall Officials: Ayana Jordan, MD, PhD., Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - Beulah Heights First Pentecostal Church, New Haven, Connecticut
  - Dixwell Ave Congregational United Church of Christ, New Haven, Connecticut
  - The Substance Abuse Training Unit (SATU), New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No